CLINICAL TRIAL: NCT05692284
Title: The Effect of Self-Care Insufficiency Care Model and Mobile Application Supported Care on Symptoms and Quality of Life of Gastrointestinal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yasemin Ciraci Yasar, Research Assistant, Ataturk University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtaturkU-NRS-YCY-01
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Nursing Care for Gastrointestinal Cancer Patients
Keywords: nursing care; mobil application; Orem's theory; self care

STUDY DESIGN:
Intervention Model Description: In the study, 60 individuals, including 1 experimental and 1 control group, were included in the study.
Who Masked: Participant
Masking Description: The patients in the control and intervention groups did not know which group they belonged to, only the researcher knew who was in which group, and the study was continued single-blindly by providing blinding in this way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine care group (Other): Routine clinic nursing care in hospital, no follow-up after discharge.
  Interventions: Other: routine care group
- Care in accordance with Orem's theory group (Experimental): care in accordance with Orem's theory in the hospital process and follow-up with a mobile application designed according to Orem's theory after discharge
  Interventions: Other: Care in accordance with Orem's theory group

INTERVENTIONS:
Other: routine care group — Firstly, informed consent was obtained from the patients in the control group, a pre-test was applied with the existing data collection methods, and routine nursing care continued. At the end of the 6-week follow-up period, the data collection process was ended with the post-test application.
  Arms: routine care group
Other: Care in accordance with Orem's theory group — Firstly, informed consent was obtained from the Intervention group, for which the pre-test was applied, and then care was given during their stay in the hospital in accordance with Orem's theory. This care was performed when the patient came to each chemotherapy cycle. After discharge, patient follow-up and care continued with the mobile application designed with Orem's theory, which will ensure the continuity of this care given in the clinic. At the end of the 6-week follow-up period, the data collection process was ended with the post-test application.
  Arms: Care in accordance with Orem's theory group

SUMMARY:
Remarkably, the incidence of gastrointestinal cancer cases among cancer types is increasing. Gastrointestinal cancers are one of the 10 most common cancer types in the World. This increase worldwide is remarkable, especially due to the increase in urbanization, consumption of foods rich in animal fat, insufficient dietary fiber intake and lifestyle changes. Cytotoxic therapy, which is used in the treatment of malignant diseases, can cause serious complications in gastrointestinal cancer, distinguishing it from other types of cancer. In addition, patients experience symptoms such as nausea-vomiting, mucositis, diarrhea, and constipation much more severely due to the direct effects of these agents on the gastrointestinal system. For this reason, patients' compliance with the treatment process and their quality of life are seriously affected, and patients have difficulties especially in meeting their self-care needs.

DETAILED DESCRIPTION:
Remarkably, the incidence of gastrointestinal cancer cases among cancer types is increasing. Gastrointestinal cancers are one of the 10 most common cancer types in the World. This increase worldwide is remarkable, especially due to the increase in urbanization, consumption of foods rich in animal fat, insufficient dietary fiber intake and lifestyle changes. Cytotoxic therapy, which is used in the treatment of malignant diseases, can cause serious complications in gastrointestinal cancer, distinguishing it from other types of cancer. In addition, patients experience symptoms such as nausea-vomiting, mucositis, diarrhea, and constipation much more severely due to the direct effects of these agents on the gastrointestinal system. For this reason, patients' compliance with the treatment process and their quality of life are seriously affected, and patients have difficulties especially in meeting their self-care needs. The aim of this project is to evaluate the effects of self-care deficit care model and mobile application-supported care on symptoms and quality of life of patients with gastrointestinal cancer.

Material and method: The research was conducted as a experimental study. The universe of the research; Between Feb 2022 and Jan 2023, individuals who met the criteria for inclusion in the study who applied for home care to Erzurum Atatürk University Research Hospital Oncology Clinic with the diagnosis of gastrointestinal cancer. The sample size for the research was determined by power analysis. In the power analysis, it was determined that a total of 52 people should be reached in order to reach the 95% confidence level at the 0.05 significance level and 80% power at the p<0.05 significance level. Considering that there may be data losses in the study, it was decided to reach 60 people, 15% more than the sample. The patients included in the study were determined as intervention (n=30) and control (n=30). During the data collection process, 4 patients, 1 in the control group and 3 in the experimental group, died and the study was completed with the results of 29 control and 27 intervention group patients. "Patient Description Form" from the intervention and control group to determine the current physical and psychological self-care needs of patients with gastrointestinal cancer, "Edmonton Symptom Assesment Scale" physical symptoms experienced by patients, and "Quality of Life Scale" for psychological symptoms and the "Self care ability scale" for self care ability was used to collect information. Permissions for use were obtained for each of the scales. In the analysis of data; percentile distribution, chi-square, Fisher-Freeman- Halton Exact test, t-test in independent groups, Repeated Measures ANOVA Test, Friedman Test, One Way ANOVA test, Kruskall Wallis test, and post hoc analyzes (Bonferroni, Games Howell, Dunn) were used.

In the intervention group, symptoms on the ESAS improved significantly. The EORTC QLQC30 functionality and symptom sub-dimensions improved significantly. In the control group, the severity of symptoms increased and quality of life decreased compared to baseline measurements. While self-care competence increased significantly in the experimental group, there was no change in the control group. The need to develop "common language, common care" practices in oncology clinics, accompanied by an evidence-based guide, is also a priority in patient care. The results of this study showed that mobile app-supported Orem's care can effective on patients' symptoms, and self care ability.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Being diagnosed with gastrointestinal cancer
* Being receiving chemotherapy treatment and having information about the disease
* Getting a score of 120 or less in the Self-Care Strength Scale pre-test.
* Not having a physical illness or cognitive disability that prevents participation in the -research and not having a psychiatric illness diagnosis
* Having an Android phone and the ability to use it
* Not having sensory loss related to vision and hearing
* Being open to communication and cooperation

Exclusion Criteria:

* Patients who did not meet the inclusion criteria and were not volunteers were not included in the sample;
* Asking to leave the study
* Worsening of general condition/Death
* Change of treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Patient Identification Form | 6 weeks
  Personal information form prepared by the researcher in line with the relevant literature; It consists of 20 questions that include socio-demographic characteristics such as age, gender, social security, educational status, disease-related features such as drugs used and duration of the disease.

SECONDARY OUTCOMES:
Edmonton Symptom Assesment Scale (ESAS) | 6 weeks
  ESAS was developed to evaluate nine common symptoms in cancer patients. These symptoms are; pain, fatigue, nausea, sadness, anxiety, insomnia, loss of appetite, well-being, shortness of breath and other problems. The severity of each symptom is assessed by numerical numbers from 0 to 10. A score of 0 indicates that there is no symptom, and a score of 10 indicates that the symptom is felt very severely, and the severity of the symptom increases from 0 to 10.
EORTC QLQC30 Quality of Life Scale | 6 weeks
  The EORTC-QLQ-C30 Quality of Life Scale is a scale developed by EORTC and includes three sub-headings of general well-being, functional difficulties, symptom control, and 30 questions. None: 1, Slightly: 2, Quite: 3, or A lot: 4 points.
SELF CARE ABILITY SCALE | 6 weeks
  The Self-Care Ability Scale is used to determine the ability of individuals to take care of themselves. A high total score from the Self-Care Scale indicates that the patients are independent and sufficient in performing their self-care. There are 35 statements in the Turkish form and each statement is evaluated with scores ranging from 0 to 4. They are listed as 0 (does not describe me at all), 1 (does not describe me very well), 2 (no idea), 3 (describes me a little), 4 (describes me a lot). Eight statements in the scale (3, 6, 9, 13, 19, 22, 26 and 31) are evaluated as negative and scoring is reversed. Evaluation is made out of a total of 140 points. Below 82 points is considered as low, 82-120 points as medium, above 120 points as high.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No